CLINICAL TRIAL: NCT04904328
Title: A Proof of Concept Clinical Investigation Designed to Evaluate the Performance of Lumishade® Lens With Frame in Alleviating the Symptoms of Photosensitive Migraine.
Brief Title: A Proof of Concept Alleviating the Symptoms of Photosensitive Migraine.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mitsui Chemicals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LUMIS001; ID: 273901 (Other: IRAS)
Record Dates: First submitted 2021-05-18; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Migraine
Keywords: Migraine; Aura; Photosensitivity; Wavelength; Lens; Glasses
MeSH Terms: conditions — Migraine Disorders; Epilepsy; Photosensitivity Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumishade® active lens (Active Comparator): Treatment of photosensitive migraine with a Lumishade® active device.
  Interventions: Device: Lumishade® Active Lens
- Lumishade® sham lens (Sham Comparator): Treatment of photosensitive migraine with a Lumishade® sham device.
  Interventions: Device: Lumishade® Sham Lens

INTERVENTIONS:
Device: Lumishade® Active Lens — Migraine episodes are often triggered or exacerbated by environmental factors, particularly light. Active lens has been designed by blocking particular range of wavelength and hypothetically alleviate symptoms of migraine and thus either treat or prevent migraine headaches from occurring.
  (Note, we are reluctant to write any further information around the devices on this public record while the study is active to ensure we maintain the blind of the trial.)
  Arms: Lumishade® active lens
Device: Lumishade® Sham Lens — Lumishade® Sham lens has been designed as inactive and not blocking particular range of wavelength. Thus, it will not alleviate or prevent symptoms of migraine.
  (Note, we are reluctant to write any further information around the devices on this public record while the study is active to ensure we maintain the blind of the trial.)
  Arms: Lumishade® sham lens

SUMMARY:
This proof of concept clinical study will investigate the efficacy of active lens with frame in alleviating the symptoms of migraine which are caused by photosensitivity.

The spectacles cut out blue light wavelength and hypothetically alleviate symptoms of migraine and thus either treat or prevent migraine headaches from occurring.

DETAILED DESCRIPTION:
Patients will be randomised to one of two groups:

Group 1

1. Patients wear sham glasses for 4 weeks
2. Patients have 1 week's washout
3. Patients wear active glasses for 4 weeks

   Group 2
4. Patients wear active glasses for 4 weeks
5. Patients have 1 week's washout
6. Patients wear sham glasses for 4 weeks

The study will aim to determine whether wearing the active lens successfully reduces the symptoms of migraine, compared to wearing sham lens.

Assuming a fairly conservative SD in the primary endpoint of 8 points, a total of 56 participants would be required to have 90% power to detect a minimum clinically significant difference of 5 points in a two-sample t-test. Allowing for a 20% drop-out rate, 70 participants would need to be recruited.

Patients will be in the trial for a total of 13 weeks (4 week run-in, two 4 week periods, with 1 week washout in between).

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old
2. Diagnosis of migraine before the age of 50, confirmed though screening consultation with the patient
3. Willing and able to provide written informed consent
4. Willing to comply with study assessment schedule and patient diary entry
5. Diagnosis of migraine, with or without aura based on the following primary headache characteristics (based on the Revised International Headache Society criteria for migraine headache)

   1. At least 5 attacks fulfilling criteria B-D
   2. Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)
   3. Headache has at least two of the following characteristics:

   i. unilateral location ii. pulsating quality iii. moderate or severe pain intensity iv. aggravation by or causing avoidance of routine physical activity (e.g., walking or climbing stairs) d. During headache at least one of the following: i. nausea and/or vomiting ii. photophobia and phonophobia e. Not attributed to another disorder
6. Migraine associated with photophobia i.e. either photic hypersensitivity or photic allodynia or inter-ictal photophobia or migraine triggered by light according to patient or a combination of these 4 factors
7. No expected changes of headache preventative medications after enrolment

Exclusion Criteria:

1. Patients with other light sensitive conditions, such as iritis or retinal disease.
2. Patients who have less than 4 headache days per month
3. Patients who have daily headaches.
4. Pregnant or nursing
5. History of cluster headache or hemiplegic migraine
6. Evidence of seizure or major psychiatric disorder
7. Score of 19 or higher on the BDI
8. Active chronic pain syndrome
9. Cardiac or hepatic disease
10. Have taken any investigational medication within 12 weeks before randomization, or are scheduled to receive an investigational drug
11. Have received Botox injections for any purpose in the head or face region within 3 months of trial onset or scheduled to receive such treatment during the trial
12. Medication overuse as per the revised ICHD-3 IHS criteria
13. Medications that can affect light perception like ethambutol, hydroxychloroquine or amiodarone or any other according to the opinion of the investigator
14. Patients requiring prescription/reading glasses
15. Patients who have not responded to three or more migraine preventive drugs
16. Patients who have a diagnosed neurological disorder that may influence the study according to the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2022-01-04 (Estimated); Study Completion 2022-04-04 (Estimated)

PRIMARY OUTCOMES:
Headache Impact Test 6 | up to 13 weeks for each patients participation
  The primary endpoint is the change in Headache Impact Test (HIT-6) score from end of run-in (Baseline) to end of treatment period following 4 weeks of treatment. The HIT 6 questionnaire is a licensed questionnaire with standardised calculations to assess the responses to the questions in the questionnaire.

SECONDARY OUTCOMES:
Patient diary | up to 13 weeks for each patients participation
  A headache diary. A headache diary serves to:
  * Monitor the frequency, duration and severity of your headaches over time
  * Identify patterns that may help determine triggers and improve treatment
  * Track medication use and response
  * Maintain long term records of what has worked and what has not

IPD SHARING:
Plan to Share IPD: No